CLINICAL TRIAL: NCT00769145
Title: Ranibizumab for the Inhibition of Neovascularization in the Cornea Following Corneal Transplant Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sonia Yoo, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20071015
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Corneal Neovascularization
Keywords: Corneal neovascularization; Ranibizumab; Corneal transplantation
MeSH Terms: conditions — Corneal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental): Patients to receive two injections of 0.5 mg ranibizumab subconjunctivally
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5mg subconjunctival dose of ranibizumab 3 days prior to corneal transplantation and at the time of corneal transplantation (total 2 injections).
  Other Names: Lucentis

SUMMARY:
The primary purpose of this trial is to evaluate the safety and tolerability of ranibizumab given via subconjunctival injection in patients undergoing corneal transplantation.

DETAILED DESCRIPTION:
As a secondary objective, this study also aims to establish the corneal and anterior chamber concentration of ranibizumab when delivered subconjunctivally at the limbus in patients undergoing corneal transplantation. The effects of ranibizumab on corneal epithelial healing will be examined following adjunctive use in corneal transplantation. Finally, clinical characteristics including recurrent corneal neovascularization will be studied.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Patient related considerations
* All patients of both genders will be considered for enrollment.
* Disease related considerations
* Patients meeting accepted criteria for undergoing corneal transplantation will be considered if peripheral corneal neovascularization exists in 2 or more contiguous clock hours

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test)
* Women seeking to become pregnant
* Lactating women
* Prior enrollment in the study
* Prior glaucoma surgery in the region of the corneal neovascularization
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary purpose of this trial is to evaluate the safety and tolerability of ranibizumab given via subconjunctival injection in patients undergoing corneal transplantation. | 2 years

SECONDARY OUTCOMES:
This study also aims to establish the corneal and anterior chamber concentration of ranibizumab when delivered subconjunctivally. The effects of ranibizumab on corneal epithelial healing and prevention of recurrent neovascularization will be examined. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Yoo, MD, Principal Investigator — Bascom Palmer Eye Institute
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States